CLINICAL TRIAL: NCT01693679
Title: Telbivudine Renoprotective Effect in Patients With HBV-related Liver Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shao-quan Zhang (Other)
Responsible Party: Sponsor-Investigator, Shao-quan Zhang, Department of Infectious Diseases, The Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telbivudine
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: HBV-related Liver Cirrhosis
Keywords: Tebivudine eGFR non-Tebivudine
MeSH Terms: interventions — Telbivudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- antiviral drug (Experimental): Telbivudine team,Telbivudine,600mg/d,oral,60 patients. non-Tebivudine team,Lamivudine,100mg/d,oral,20 patients.Adefovir,10mg/d,oral,20 patients.Enecavir,0.5mg/d,oral,20 patients.
  Interventions: Drug: Telbivudine, Lamivudine, Adefovir ,Enecavir

INTERVENTIONS:
Drug: Telbivudine, Lamivudine, Adefovir ,Enecavir — investigational Telbivudine,600mg,daily,oral.comparator Lamivudine,100mg daily, oral,Adefovir,10mg,daily,oral,Enecavir,0.5mg,daily,oral.
  Other Names: no.

SUMMARY:
• To estimate renoprotective efficacy of Telbivudine treated patients with HBV-related liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

* Aged between 18-75 years (inclusive).
* Male or female.
* Subjects with positive HBsAg for more than 6 months and anti-HBs negative regardless of HBeAg status , HBV DNA ≥2×103 IU/ml
* Subjects with HBV-related liver cirrhosis, including compensated cirrhosis and decompensated, but only Child-Pugh A or B.
* The ablility to understand and sign a written informed consent prior to any study related procedure and comply with the requirements of the study.

Exclusion Criteria:

* Subjects meeting any of the following criteria must not be enrolled in the study

  * Subjects with non-HBV cirrhosis
  * Co-infection with HAV/HCV/HDV/ HIV
  * Subjects who take nucleosides within 6 months
  * Kidney injury due to non-HBV factors
  * Inability to comply with study requirements as determined by the study investigator
  * Patients with very low GFR, who may need dialysis or renal transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in glomerular filtration rate and Serum creatinine at 96 weeks | May 2014
  No.

SECONDARY OUTCOMES:
Change from Baseline in ALT normalization rate,• The rate of complications,• Percentage of participants with HBeAg loss & HBeAg seroconversion and Percentage of subjects achieving HBV DNA<300copies/mL at96 weeks | May 2014
  No.